CLINICAL TRIAL: NCT03868254
Title: XEN 45 Gel Stent: Long Term Performance and Safety Assessment (XEN LT)
Brief Title: Chart Review of XEN 45 Gel Stent: Long Term Performance and Safety Assessment (XEN LT)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: CMO-MA-EYE-0590
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Implant: Chart review was conducted in participants with open angle glaucoma who underwent placement of the implant XEN 45 Gel Stent as a standalone procedure from 1 January 2014 to 1 October 2015. For each eye selected, all retrospective data available from baseline (day when decision was made to implant XEN 45 Gel Stent) until the last visit was extracted from existing medical records.
  Interventions: Device: XEN Group
- Implant + Phaco: Chart review was conducted in participants with open angle glaucoma who underwent placement of the implant XEN 45 Gel Stent in combination with phacoemulsification (Phaco) from 1 January 2014 to 1 October 2015. For each eye selected, all retrospective data available from baseline (day when decision was made to implant XEN 45 Gel Stent) until the last visit was extracted from existing medical records.
  Interventions: Procedure: Phacoemulsification

INTERVENTIONS:
Device: XEN Group — Chart review was conducted in participants with open angle glaucoma who underwent placement of the implant XEN 45 Gel Stent as a standalone procedure from 1 January 2014 to 1 October 2015.
  Groups: Implant
Procedure: Phacoemulsification — Chart review was conducted in participants with open angle glaucoma who underwent placement of the implant XEN 45 Gel Stent in combination with phacoemulsification (Phaco) from 1 January 2014 to 1 October 2015.
  Groups: Implant + Phaco

SUMMARY:
A retrospective, non-interventional, observational, multi-center, chart review study to be conducted in participants who underwent placement of the XEN 45 Gel Stent as a standalone procedure or in combination with phacoemulsification from 1 January 2014 to 1 October 2015.

ELIGIBILITY:
Inclusion Criteria:

* Eye treated with XEN 45 Gel Stent for primary open angle glaucoma as a standalone procedure or in combination with phacoemulsification
* XEN 45 Gel Stent was implanted between 1 January 2014 and 1 October 2015

Exclusion Criteria

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participant eyes that underwent XEN 45 Gel Stent implantation from 1 January 2014 until 1 October 2015.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mini Balaram, MD, Study Director — Allergan
Locations (1):
- Clinical Trials Registry Team, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Implant | Implant + Phaco
Started | 98; 116 Eyes | 76; 96 Eyes
Completed | 98; 116 Eyes | 76; 96 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Population: Effectiveness Population consisted of all eligible participant eyes. In instances when a participant contributed both eyes in study eye that received XEN 45 Gel implant first was selected (primary eye).
Units Other Than Participants: eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Implant | Implant + Phaco | Total
Number analyzed (Participants) | 98 | 76 | 174
Number analyzed (eyes) | 98 | 76 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.40 (12.193) | 75.95 (7.107) | 72.26 (10.764)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 39 | 91
  Male | 46 | 37 | 83
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Caucasian | 91 | 75 | 166
  Latin American | 1 | 1 | 2
  Asian | 4 | 0 | 4
  Unknown | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Intraocular Pressure (IOP) to 36 Months After Implantation
Description: IOP is a measurement of the fluid pressure inside the eye. A negative change from Baseline indicates an improvement.
Time Frame: Baseline (Day decision was made to implant XEN 45 Gel Stent) to 36 months after implantation
Population: Participants from effectiveness population, all eligible participant eyes with data available at Baseline.In instances when a participant contributed both eyes, eye that received XEN45Gel implant first was selected(primary eye).Analysis included 1 eye for each participant.Number analyzed:number of participants and eyes analyzed at given timepoint.
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: eyes
Arm/Group | Implant | Implant + Phaco
Number analyzed (Participants) | 90 | 73
Number analyzed (eyes) | 90 | 73
mm Hg
  Baseline | 21.03 (4.638) | 20.21 (5.640)
  Change from Baseline to Month 36: number analyzed (Participants) | 46 | 30
  Change from Baseline to Month 36: number analyzed (eyes) | 46 | 30
  Change from Baseline to Month 36 | -6.42 (5.655) | -6.73 (7.620)
Statistical Analysis 1: Comparison: Implant; Test type: Other; p < .0001, Paired t-test
Statistical Analysis 2: Comparison: Implant + Phaco; Test type: Other; p < .0001, Paired t-test

2. Primary Outcome: Change From Baseline in the Number of Topical IOP-lowering Medications 36 Months After Implantation
Description: IOP-lowering medications included Beta blocking agents, Carbonic anhydrase inhibitors, Parasympathomimetics, Prostaglandin analogues, and Sympathomimetics in glaucoma therapy.
Time Frame: Baseline (Day decision was made to implant XEN 45 Gel Stent) to 36 months after implantation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: medications
Units Other Than Participants: eyes
Arm/Group | Implant | Implant + Phaco
Number analyzed (Participants) | 90 | 73
Number analyzed (eyes) | 90 | 73
medications
  Baseline | 2.6 (0.98) | 2.4 (1.02)
  Change from Baseline to Month 36: number analyzed (Participants) | 46 | 30
  Change from Baseline to Month 36: number analyzed (eyes) | 46 | 30
  Change from Baseline to Month 36 | -1.6 (1.49) | -1.2 (1.52)
Statistical Analysis 1: Comparison: Implant; Test type: Other; p < .0001, Paired t-test
Statistical Analysis 2: Comparison: Implant + Phaco; Test type: Other; p = 0.0001, Paired t-test

3. Secondary Outcome: Change From Baseline in Mean IOP to 48 Months After Implantation
Description: IOP is a measurement of the fluid pressure inside the eye. A negative change from Baseline indicates an improvement.
Time Frame: Baseline (Day decision was made to implant XEN 45 Gel Stent) to 48 months after implantation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Units Other Than Participants: eyes
Arm/Group | Implant | Implant + Phaco
Number analyzed (Participants) | 90 | 73
Number analyzed (eyes) | 90 | 73
mm Hg
  Baseline | 21.03 (4.638) | 20.21 (5.640)
  Change from Baseline to Month 48: number analyzed (Participants) | 12 | 15
  Change from Baseline to Month 48: number analyzed (eyes) | 12 | 15
  Change from Baseline to Month 48 | -5.46 (4.998) | -5.27 (5.298)
Statistical Analysis 1: Comparison: Implant; Test type: Other; p = 0.0030, Paired t-test
Statistical Analysis 2: Comparison: Implant + Phaco; Test type: Other; p = 0.0018, Paired t-test

4. Secondary Outcome: Change From Baseline in the Number of Topical IOP-lowering Medications 48 Months After Implantation
Description: as for outcome 2
Time Frame: Baseline (Day decision was made to implant XEN 45 Gel Stent) to 48 months after implantation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: medications
Units Other Than Participants: eyes
Arm/Group | Implant | Implant + Phaco
Number analyzed (Participants) | 90 | 73
Number analyzed (eyes) | 90 | 73
medications
  Baseline | 2.6 (0.98) | 2.4 (1.02)
  Change from Baseline to Month 48: number analyzed (Participants) | 12 | 15
  Change from Baseline to Month 48: number analyzed (eyes) | 12 | 15
  Change from Baseline to Month 48 | -1.1 (1.08) | -0.8 (1.42)
Statistical Analysis 1: Comparison: Implant; Test type: Other; p = 0.0053, Paired t-test
Statistical Analysis 2: Comparison: Implant + Phaco; Test type: Other; p = 0.0472, Paired t-test

5. Secondary Outcome: Percentage of Eyes Achieving Qualified Success at Month 36
Description: Qualified success of implantation of the XEN 45 Gel Stent is defined as ≥20% reduction in IOP from medicated baseline with no SSI for glaucoma and no clinical hypotony while staying on the same number or fewer topical IOP-lowering medications than at Baseline.
Time Frame: Baseline (Day decision was made to implant XEN 45 Gel Stent), Month 36
Population: Participants from effectiveness population, consisting of all eligible participants eyes, with data available for analyses. In instances when a participant contributed both eyes in the study, the eye that received XEN 45 Gel implant first was selected (primary eye). Analysis included one eye for each participant.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Implant | Implant + Phaco
Number analyzed (Participants) | 46 | 30
Number analyzed (eyes) | 46 | 30
percentage of eyes | 23.9 | 40.0

6. Secondary Outcome: Percentage of Eyes Achieving Qualified Success at Month 48
Description: as for outcome 5
Time Frame: Baseline (Day decision was made to implant XEN 45 Gel Stent), Month 48
Population: as for outcome 5
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Implant | Implant + Phaco
Number analyzed (Participants) | 12 | 15
Number analyzed (eyes) | 12 | 15
percentage of eyes | 25.0 | 33.3

7. Secondary Outcome: Percentage of Eyes Achieving Complete Success at Month 36
Description: Complete success of implantation of the XEN 45 Gel Stent is defined as ≥20% reduction in IOP from Baseline with no SSI for glaucoma and no clinical hypotony while taking no topical IOP-lowering medications.
Time Frame: Baseline (Day decision was made to implant XEN 45 Gel Stent), Month 36
Population: as for outcome 5
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Implant | Implant + Phaco
Number analyzed (Participants) | 46 | 30
Number analyzed (eyes) | 46 | 30
percentage of eyes | 45.7 | 20.0

8. Secondary Outcome: Percentage of Eyes Achieving Complete Success at Month 48
Description: as for outcome 7
Time Frame: Baseline (Day decision was made to implant XEN 45 Gel Stent), Month 48
Population: as for outcome 5
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Implant | Implant + Phaco
Number analyzed (Participants) | 12 | 15
Number analyzed (eyes) | 12 | 15
percentage of eyes | 33.3 | 20.0

9. Secondary Outcome: Percentage of Eyes With Adverse Events of Special Interest (AESIs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with use of a drug whether or not it is considered related to drug. AESI include: Glaucoma, defined as damage to optic nerve with progressive vision loss, Intraocular hypertension, defined as IOP without meeting criteria for glaucoma, Hypotony, defined as low IOP ≤5 mmHg, Cataract or lens opacities, Ocular bleeding or hemorrhage, Retinal detachment, tear or hole, Vitreous detachment, Infection vs. Non-infection related Ocular inflammation, Significant vitreous loss, Mechanical failure of device and implant misplacement, Implant dislocation. Data of AESIs are presented based on eyes for this outcome measure.
Time Frame: Baseline (Day decision was made to implant XEN 45 Gel Stent) to approximately 51 Months
Population: Safety Population consisted of all eligible participant eyes in the study population. For participants implanted bilaterally, both eyes were included for analysis if both met the eligibility criteria.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Implant | Implant + Phaco
Number analyzed (Participants) | 98 | 76
Number analyzed (eyes) | 116 | 96
percentage of eyes | 18.1 | 10.4

ADVERSE EVENTS:
Time Frame: Baseline (Day decision was made to implant XEN 45 Gel Stent) to approximately 51 Months
Description: Only AESIs were collected for this study.
Arm/Group | Implant | Implant + Phaco
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/76
Serious Adverse Events (participants affected / at risk) | 2/98 | 0/76
Other Adverse Events (participants affected / at risk) | 0/98 | 0/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Implant (N=98) | Implant + Phaco (N=76)
Bleb leak (Eye disorders) | 1 | 0
Endophthalmitis (Eye disorders) | 1 | 0
Persistent Hypotony (Eye disorders) | 1 | 0
Clinical Hypotony (Eye disorders) | 1 | 0
Anterior chamber defects (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT03868254/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT03868254/SAP_001.pdf